CLINICAL TRIAL: NCT05008640
Title: TrueLoo™: Determining the Feasibility of an Electronic Bowel Movement and Urinary Event Log Via In Situ Categorization of Physical Properties of Stool and Urine
Brief Title: Creation of an E-toileting Log Through Classification of the Physical Properties of Stool and Urine Using TrueLoo™
Status: Completed | Type: Observational
Sponsor: Toi Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20191822; 20191822 (Other: WCG IRB (IRB #)); TLSD-001 (Other: WCG IRB (Protocol #))
Record Dates: First submitted 2021-07-14; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Urinary Tract Infections; Infectious Diarrhea; Clostridium Difficile Infection; Gastrointestinal Disease; GastroIntestinal Bleeding
Keywords: Geriatric; Gastroenterology; Urinary
MeSH Terms: conditions — Urinary Tract Infections; Dysentery; Clostridium Infections; Gastrointestinal Diseases; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group (all subjects): All subjects belonged to the same study group, regardless of symptoms, disease diagnosis or state. Furthermore, there was no stratification of the population by sex, age, race or disease severity.
  Interventions: Device: TrueLoo™

INTERVENTIONS:
Device: TrueLoo™ — TrueLoo™ is an Internet-connected, smart toilet seat that uses computer vision technology to log and capture daily bowel movements and urinations. This data is then categorized by physical excreta characteristics to train and develop machine learning algorithms that are intended to eventually identify significant changes in stool and urine in real-time.

SUMMARY:
The purpose of this study is to assess the feasibility of TrueLoo™, an Internet-connected smart toilet seat, in accurately monitoring and logging bowel movements and urinations of residents in senior living facilities across Northern California.

DETAILED DESCRIPTION:
The logging and monitoring of bowel movements and urinary events is an important aspect of preventative care for residents in senior living facilities, providing early warning signs for conditions that may otherwise cause complications if dealt with reactively. However, this information is sporadically collected - if at all - and subjectively interpreted by caregivers, leading to inconsistencies and unreliable data. Toi Labs, Inc. has created TrueLoo™, an Internet-connected toilet seat, as a solution to these issues. TrueLoo™ acquires time-lapse images of a bowel movement or urinary event automatically and under controlled conditions. Residents enrolled in the current study will have a TrueLoo™ installed in their private bathroom, through which all bowel movements and urinary events will be tracked, anonymously, privately, and securely. As a result, an electronic bowel movement and urinary event log for each enrolled resident will be generated. Given sufficient data, the TrueLoo™ system will complete such electronic logs automatically, identify points in time where particular enrolled residents may have experienced anomalous toileting patterns, and determine the relevance of such events through targeted health history and urine sampling.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to participate and provide consent for the study;
* Must be a male or female, aged 55 or older;
* Must be a resident of a senior living facility;
* Must have regular access to a TrueLoo™.

Exclusion Criteria:

* Candidates who are unwilling or unable to accept the requirements associated with installing TrueLoo™ in their residence, including power and Wi-Fi connectivity;
* Candidates who use certain types of toileting assistance devices that at this time are not compatible with TrueLoo™ (e.g., padded toilet seat risers).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population was comprised of subjects that belong to the same study group, regardless of symptoms, disease diagnosis or state. Furthermore, there was no stratification of the population by sex, age, race or disease severity.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Bowel movement and urinary event dataset creation | Week 16 - 30
  Number of urinations and bowel movements exhibited from each participant during the study period, as observed by TrueLoo™ image analysis.

SECONDARY OUTCOMES:
Comparison with current methodologies | Week 16 - 30
  Error rate of bowel movement and urinary event tracking from current caregiver-reported and self-reported methods.

OTHER OUTCOMES:
Identification of anomalous toileting patterns in TrueLoo™ data | Week 16 - 30
  Number of bowel movement and urinary event anomalies observed by TrueLoo™; ad-hoc health history collection and urine sampling will determine the relevance of these events.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Cristman, PhD, MS, BS, Principal Investigator — Toi Labs, Inc.
Locations (6):
- United States (6):
  - Carlton Senior Living (Concord), Concord, California
  - Carlton Senior Living (Davis), Davis, California
  - Carlton Senior Living (Elk Grove), Elk Grove, California
  - Eskaton Village Carmichael, Sacramento, California
  - Eskaton Lodge Cameron Park, Sacramento, California
  - Masonic Homes, Union City, California

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT05008640/ICF_000.pdf